CLINICAL TRIAL: NCT00317928
Title: Efficacy of Metformin in PCOS: Metabolic and Hormonal Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Regional Hospital Holstebro (Other); Aarhus University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 160350-1
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2001-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Metformin; Metabolic Syndrome; Hyperandrogenism; Ovulation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome; Hyperandrogenism | interventions — Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Hypothesis: Metformin treatment normalises hormone values and metabolic parameters in women with PCOS. Ovulation is restored and bleeding periods become regular.

Fifty women with PCOS (Rotterdam criteria) are randomised to either placebo or metformin for 6 months. After a wash-out period of 3 months, the opposite treatment is given for another 6 months. Measurements are performed before ech treatment period, every second month during treatment and after completing treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS
* Age 20 - 45

Exclusion Criteria:Diabetes

* Diabetes
* Hormonal treatment
* Pregnancy, lactation
* Periclimacteric

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 2001-08; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Trolle, MD, Principal Investigator — Skejby University Hospital, Aarhus, Denmark